CLINICAL TRIAL: NCT05716737
Title: Exploring Radiotherapy of Temporomandibular Joint Arthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Cora Waldstein, Principal Investigator, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMJRT1107/2023
Record Dates: First submitted 2023-01-30; First posted 2023-02-08 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Arthritis of Temporomandibular Joint
MeSH Terms: interventions — Radiation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TMJ RT (Experimental): Patients receiving irradiation to the TMJ
  Interventions: Radiation: Irradiation

INTERVENTIONS:
Radiation: Irradiation — 3 Gy in 6 fractions to the TMJ, every other day, LINAC based

SUMMARY:
With this pilot study, the acute side effects and potential pain relieve after radiotherapy (RT) of the temporomandibular joint (TMJ) are prospectively recorded.

For this purpose, the symptoms of the jaw joint arthrosis/arthritis are recorded using a symptom-oriented questionnaire and the numeric rating scale for pain assessment.

Furthermore, it is examined whether the irradiation is feasible.

ELIGIBILITY:
Inclusion Criteria:

* TMJ arthritis
* diagnosed by a surgeon for oral and maxillofacial surgery or a dentist

Exclusion Criteria:

* Previous irradiation in the TMJ area
* Age below 50 years

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-07-07 (Actual); Primary Completion 2024-07-07 (Actual); Study Completion 2027-07-07 (Estimated)

PRIMARY OUTCOMES:
therapeutic effect | Before, directly after treatment and after 3, 6 9 and 12 months
  Pain, Numeric rating scale (0-10, 0=no pain, 10=maximum pain)

SECONDARY OUTCOMES:
Other temporomandibular joint conditions | Before, directly after treatment and after 3, 6 9 and 12 months
  Questionnaire (covering the condition of the temporomandibular joint and masticatory muscles, Version: 12.03.2018 (FB II) of the University of Leipzig)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No